CLINICAL TRIAL: NCT01926002
Title: A Multicenter Randomized Clinical Trial to Study the Effects of Single Doses of MK-8351 on the Early Asthmatic Response to a Lung Allergen Challenge
Brief Title: A Single-Dose Study of MK-8351 in a Lung Allergen Challenge (MK-8351-003)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 8351-003; MK-8351-003 (Other: Merck Study Number)
Record Dates: First submitted 2013-08-16; First posted 2013-08-20 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low-Dose MK-8351 (Experimental): Low-dose MK-8351 administered as single inhaled dose.
  Interventions: Drug: Low-Dose MK-8351
- High-Dose MK-8351 (Experimental): High-dose MK-8351 administered as a single inhaled dose.
  Interventions: Drug: High-Dose MK-8351
- Placebo to MK-8351 (Placebo Comparator): Matching placebo to low-dose or high-dose MK-8351 administered as a single inhaled dose.
  Interventions: Drug: Placebo to MK-8351

INTERVENTIONS:
Drug: Low-Dose MK-8351 — Single administration of low-dose MK-8351.
  Arms: Low-Dose MK-8351
Drug: High-Dose MK-8351 — High-Dose MK-8351 administered as a single inhaled dose.
  Arms: High-Dose MK-8351
Drug: Placebo to MK-8351 — Single-Dose Matching placebo to high-dose or low-dose MK-8351.
  Arms: Placebo to MK-8351

SUMMARY:
The primary hypothesis of the study is single doses of MK-8351 will reduce the baseline early asthmatic response (EAR) as assessed by area under the curve from 0-3 hours (AUC0-3hr) of forced expiratory volume (FEV1) when compared to placebo.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, 4-period study. Eligible patients will undergo a single-blind phase in Period 1, followed by 3 periods during which they will receive low-dose MK-8351, high-dose MK-8351, or matching placebo as a single dose in a random sequence crossover study design.

ELIGIBILITY:
Inclusion Criteria:

* Females of non-childbearing potential (at least 1 year post-menopausal, post-hysterectomy, post-oophorectomy, or with tubal ligation);
* Males with a female partner of childbearing potential must agree to use a medically acceptable method of contraception during and up to 120 days after the last dose of study medication;
* Body Mass Index (BMI) >=17 kg/m^2 and <=33 kg/m^2
* Non-smoker and non-user of nicotine or nicotine-containing products for at least 6 months prior to enrollment;
* History of allergen-induced asthma for at least 6 months prior to enrollment;
* Able to perform reproducible pulmonary function testing;
* Positive methacholine challenge test prior to receiving study medication;
* Allergic response to house dust mite allergen or standardized cat pelt or hair allergen extract;
* Ability to tolerate sputum induction and to produce adequate sputum.

Exclusion Criteria:

* History of clinically significant disease or disorder;
* History of malignancy;
* History of significant multiple and/or severe allergies;
* History of milk or lactose allergies or intolerance;
* History of anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food;
* Positive for human immunodeficiency virus (HIV), hepatitis B surface antigen, or hepatitis C antibodies;
* History of major surgery within 3 months prior to enrollment;
* Participation in another investigational trial within 4 weeks of screening;
* Lactating females;
* Inability to refrain from, or anticipates the use of, any medication including herbal remedies during the trial period;
* History of receiving anti-immunoglobulin E (IgE) or immunotherapy;
* History of serious allergies to drug or a history of hypersensitivity to inhaled salbutamol, antihistamines, or any other potential asthma/anaphylaxis rescue medication;
* History of hospitalization for asthma-related illness within 3 months of screening;
* History of emergent care more than twice in the last 12 months for asthma-related illness;
* History of life-threatening asthma;
* Consumes >4 glasses of alcoholic beverage per day;
* Consumes >6 servings of coffee, tea, cola, energy drinks or other caffeinated beverages per day;
* History or or current use of illicit drugs within past 24 months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
AUC0-3hr of FEV1 Percent Change From Baseline | 3 Hours
Number of Participants Experiencing Adverse Events (AEs) | Up to 14 Days
Number of Participants Discontinuing Study Treatment Due to AEs | Up to 72 Hours

SECONDARY OUTCOMES:
AUC0-24h of MK-8351 | Up to 24 Hours Post-Dose
AUC0-last of MK-8351 | Up to 72 Hours Post-Dose
AUC0-∞ of MK-8351 | Up to 72 Hours Post-Dose
Maximum Plasma Concentration (Cmax) of MK-8351 | Up to 72 Hours Post-Dose
Time to Maximum Plasma Concentration (Tmax) of MK-8351 | Up to 72 Hours Post-Dose
Apparent Half-Life (t1/2) of MK-8351 | Up to 72 Hours Post-Dose